CLINICAL TRIAL: NCT00465842
Title: Protein Biomarkers for Early Detection and Prognostication in Hepatocellular Carcinoma (HCC)
Brief Title: Protein Biomarker in Hepatocellular Carcinoma
Status: Terminated | Type: Observational
Why Stopped: Loss of funding due to difficulty with recruitment and participant retention.
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Singapore Cancer Society (Other)
Responsible Party: Sponsor
Other Study IDs: JS0541; NA_00037477 (Other: JHM IRB)
Record Dates: First submitted 2007-04-23; First posted 2007-04-25 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Normal Volunteers; Hepatitis; Liver Cirrhosis; Hepatocellular Carcinoma
Keywords: Hepatitis; Liver Cirrhosis; HCC
MeSH Terms: conditions — Hepatitis; Liver Cirrhosis; Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- A - Normal Volunteers: Normal volunteers without any history of liver disease and with normal liver functions test (LFT), including total protein/Albumin, LDH, ALT, AST, GGT, total bilirubin, direct and indirect bilirubin and do not belong to group B.
  Volunteers will be screened using questionnaires. Those deemed suitable will then be asked to have the blood test done. All blood tests are done free of charge to subjects.
- B - Hepatitis B or C carriers with normal liver functions
- C - Hepatitis B or C carriers with abnormal liver functions
- D - Liver Cirrhosis: Liver cirrhosis, proven by liver biopsy or on clinical evidences, such as varices on CT scan indicative of portal hypertension.
- E - Hepatocellular Carcinoma (HCC) with Resection: HCC patients with resection.
- F - Unresectable HCC: Unresectable HCC patients with treatment
- G - Malignant HCC: HCC patients with active malignant disease and only palliative care are offered.

SUMMARY:
Hepatocellular carcinoma (HCC) is the fifth commonest cancer in the world with poor prognosis, as the annual mortality is almost equivalent to the incidence. This is mainly due to late diagnosis and co-morbid liver dysfunction. HCC is prevalent in our region than in the West due to prevalent Hepatitis B infection and carriers. At the time of diagnosis, only 10 - 20% of HCC patients are candidates for liver resection or transplantation. Almost 40-50% of patients have such poor liver function and co-morbid conditions that only supportive cares are offered. Thus the median survival time is 18-24 months for resectable disease, 6 months for unresectabe disease and 3 months for metastatic disease.

Current screening methods for HCC in high risk patients depend on alpha-fetoprotein (AFP) and ultrasound of the liver. Neither test is sensitive or specific enough for early detection. Therefore, early diagnosis with novel protein biomarkers is needed urgently and may provides hope to improve treatment outcome.

Our preliminary study in 49 HCC patients have identified several proteins such as truncated complement C3a, albumin, B2 microglobulin, may be potentially helpful in early diagnosis. We have started a large prospective and longitudinal study in July 2006, with nearly 100 patients accrued. This application is to extend and expand our current study. We aim to (i) identify and validate novel protein biomarkers for early diagnosis of HCC (ii) conduct longitudinal proteomics with most up-to-date methods to discover new biomarker for early detection and prognostication of HCC (iii) set up gene and plasma depository and clinical database for HCC in collaboration with Singapore Tissue Network.

DETAILED DESCRIPTION:
Up to 40% of HCC patients have normal AFP. Moreover, AFP can also be elevated in patients with cirrhosis or exacerbation of chronic hepatitis. Prospective studies evaluating the value of AFP in HCC surveillance have reported sensitivities of 39-64%, specificity of 76-91% and positive predictive values of 9 -32% 9-11.

Recently, a small handful of biomarkers were identified in the blood of 49 HCC patients by SELDI / MS proteomic analysis of their blood with specificity and sensitivity both at 90% 12, 13. These were truncated complement C3a, albumin, B2 microglobulin, and histidine-rich glycoprotein. In addition, insulin growth factor (IGF) and its binding protein have been shown to be novel biomarkers of HCC 14-17. A larger prospective study is necessary to validate these findings.

Other investigators have also used Surface-enhanced laser desorption / ionization time-of-flight mass spectrometry (SELDI) to study proteomics in HCC. Most of the studies included small numbers of patients and did not include independent test set or report on reproducibility most of the time. Thus, controversies continue on both the technology of SELDI and validation of the findings. Nevertheless, Ward et al reported that Kappa and Lumda immunoglobulin light chains were elevated by an average pf 50% in the serum of HCC patients (p < 0.001, sensitivity 94%, specificity 86%) with Hepatitis C related cirrhosis 18. Schwegler et al reported that SELDI-TOF MS profiling of serum can distinguish chronic Hepatitis C from HCV- related HCC with a sensitivity of 61% and a specificity of 76%. Sensitivity and specificity can be improved with the addition of AFP, des-gamma carboxyprothrombin, and GP73 19. Other reports also indicated potential marker of heat-shock protein 27 20 and complement C3a 21. However, all studies lack prospective and longitudinal follow-up with multiple serum samples from same patient. Our trial is designed to test the changes of proteomic overtime to identify the earliest possible biomarkers for HCC.

ELIGIBILITY:
Inclusion Criteria:

* Group A: Normal volunteers without any history of liver disease and with normal liver functions test (LFT), including total protein/Albumin, LDH, ALT, AST, GGT, total bilirubin, direct and indirect bilirubin and do not belong to group B. Volunteers will be screened using questionnaires. Those deemed suitable will then be asked to have the blood test done. All blood tests are done free of charge to subjects.
* Group B: Hepatitis B or C carriers with normal liver functions.
* Group C: Hepatitis B or C carriers with abnormal liver functions.
* Group D: Liver cirrhosis, proven by liver biopsy or on clinical evidences, such as varices on CT scan indicative of portal hypertension.
* Group E: HCC patients with resection.
* Group F: Unresectable HCC patients with treatment.
* Group G: HCC patients with active malignant disease and only palliative care are offered.
* Signed Informed Consent

  -≥ 18 years of age
* In this trial, diagnosis of HCC is established with either (a) known hepatitis B or C carrier, and space occupying lesion(s) in the liver and AFP > 400ng/ml or (b) cytological or histological confirmation by biopsy

Exclusion Criteria:

There is no exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: HCC patients, normal volunteers and patients with hepatitis with/without cirrhosis
Sampling Method: Non-Probability Sample
Enrollment: 211 (Actual)
Dates: Start 2006-06-20 (Actual); Primary Completion 2013-08-14 (Actual); Study Completion 2013-08-14 (Actual)

PRIMARY OUTCOMES:
Number of participants with presence of serum protein markers | Day 1
  Number of participants with truncated complement C3a, albumin, B2-microglobulin and histidine-rich glycoprotein, IGF-I, and IGF-II on first blood sample.

SECONDARY OUTCOMES:
Number of participants with hepatocellular carcinoma (HCC) with presence of protein markers. | up to 5 years
  To study the prospective and longitudinal value of these protein markers in detecting HCC by regular measurement of these proteins and follow up with routine clinical practice in high-risk patients.
Number of participants with presence of serum protein markers with resectable and unrsectable HCC. | up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Alex Chang, MD, Principal Investigator — Johns Hopkins Singapore
Locations (1):
- Johns Hopkins Singapore International Medical Center, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No